CLINICAL TRIAL: NCT05876377
Title: Use and Effectiveness of COVID-19 Vaccines Using State Vaccine Registries and Insurance Claims Data
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: C4591059; NCT05876377 (Registry Identifier: ClinicalTrials.gov)
Record Dates: First submitted 2023-05-23; First posted 2023-05-25 (Actual); Last update posted 2025-11-06 (Actual); Status verified 2025-11

CONDITIONS: SARS-CoV-2; COVID-19; Post-Acute COVID-19 Syndrome
Keywords: COVID-19 Vaccines; COVID-19 Drug Treatment
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — BNT162 Vaccine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- XBB Vaccinated (exposed): ≥14 days since receipt of Pfizer/BioNTech XBB dose prior to COVID-19 diagnosis
  Interventions: Biological: Pfizer-BioNTech COVID-19 mRNA vaccine
- XBB Unvaccinated (unexposed): Did NOT receive any XBB dose prior to COVID-19 diagnosis

INTERVENTIONS:
Biological: Pfizer-BioNTech COVID-19 mRNA vaccine — Pfizer-BioNTech COVID-19 Vaccine, is FDA licensed or authorized under Emergency Use Authorization (EUA) for active immunization to prevent coronavirus disease 2019 (COVID-19) caused by severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) in individuals 6 months of age and older.
  Other Names: Pfizer-BioNTech COVID-19 Vaccine
  Groups: XBB Vaccinated (exposed)

SUMMARY:
This study aims to use vaccination information from state vaccine registries linked with HealthVerity insurance claims for the following:

* to measure how effective the Pfizer-BioNTech vaccine is at preventing post-COVID conditions.
* to understand characteristics of patients who are receiving COVID-19 vaccines.

All patients whose information is kept unidentified in the HealthVerity database are eligible to be included for both aims of this study.

DETAILED DESCRIPTION:
The effectiveness of the COVID-19 vaccine in preventing post-COVID health conditions will be assessed (Aim 1). To do this, a retrospective cohort time-to-event design will be employed. Patients will be observed until an endpoint (post-COVID related condition) or a censoring event (BNT162b2 vaccine, Other COVID-19 vaccinations formulated for 2023-2024 respiratory season, or moderate/severe immunocompromised condition). All eligible patients must have been diagnosed with COVID-19 (index event) at cohort entry at which point vaccination status is determined. Patients then continue to contribute person-time to the time-to-event model as the study progresses. Patient data will be gathered from HealthVerity, including those enrolled in the claims database, and supplemented with information from the state's deidentified vaccine registry. Only patients eligible to receive the vaccine during the study period will be included in the analysis of post-COVID health conditions.

The second part of the study (Aim 2) will use a retrospective cohort design to examine the uptake of the vaccine in specific groups over time. Subjects will be identified through three different methods: 1) by analyzing all available dosing records in the Immunization Registry, 2) by using HealthVerity claims data based on specific calendar time periods when the vaccine was available, or 3) based on the start of pregnancy that occurs after EUA date. Patients will be followed until experiencing the vaccination under study, disenrollment, end of data or death. Vaccinations will be assessed overall and also by specific type of prior dose (mRNA vs other).

ELIGIBILITY:
Aim 1:

Inclusion Criteria:

Patients must meet all of the following criteria to be eligible for inclusion in the study:

1. Patients are required to have a COVID-19 diagnosis on or after September 25, 2023 AND
2. Patients in HealthVerity database and residing in California or Louisiana as of index date AND
3. Have ≥1 year of pharmacy and medical enrollment in HealthVerity prior to cohort entry date, allowing for up to a 30-day gap in enrollment AND
4. ≥18 years old as of index date AND
5. Have resided only in their respective state (California or Louisiana) for ≥1 year prior to index date

Exclusion Criteria:

Patients meeting any of the following criteria will not be included in the study:

1. Patients who were immunocompromised from 1 year prior to cohort entry OR
2. Patients who received any 2023-2024 XBB-adapted formulation of the COVID-19 vaccine prior to authorization (11 September 2023) OR
3. Patients who have discrepancies in sex and/or year of birth between HealthVerity claims and state immunization registry datasets OR
4. Patients who had a prior diagnosis of COVID-19 ≤180 days preceding cohort entry OR
5. Patients who received any 2023-2024 XBB-adapted formulation of the COVID-19 vaccine within 0 to 13 days prior OR 0 to 29 days post index COVID-19 diagnosis (i.e., -13 to +29 days around the index date)

Aim 2:

By Age, Bivalent (older children, adults)

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Has medical and pharmacy enrollment in HealthVerity as of August 31, 2022
2. And is age ≥12 years
3. With 6 months of continuous medical and pharmacy enrollment before calendar index date
4. And does not have evidence of moderate/severe immunocompromise as defined by CDC
5. And has evidence of ≥2 doses of COVID-19 original vaccine formulation before the calendar index date
6. And does not have original vaccine formulation within 2 months before calendar index date
7. And does not have a pregnancy start date within 9 months before or any point after calendar entry
8. And does not have discrepancies in sex and/or year of birth between HealthVerity claims and state Immunization registry datasets.

This analysis will be stratified by age: 12-17, 18-49. 50-64, 65-74, 75+, which will be measured as of August 31, 2022.

By Age, Bivalent (younger children)

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Has medical and pharmacy enrollment in HealthVerity as of 12 October 2022
2. And is age 5-11 years
3. With 6 months of continuous medical and pharmacy enrollment before calendar index date
4. And does not have evidence of moderate/severe immunocompromise as defined by CDC
5. And has evidence of ≥2 doses of COVID-19 original vaccine formulation before the calendar index date
6. And does not have original vaccine formulation within 2 months before calendar index date.

By Age, Bivalent (youngest children)

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Has medical and pharmacy enrollment in HealthVerity as of 08 December 2022
2. And is age 6 months-4 years
3. With 6 months of continuous medical and pharmacy enrollment before calendar index date
4. And does not have evidence of moderate/severe immunocompromise as defined by CDC
5. And has evidence of ≥2 doses of COVID-19 original vaccine formulation before the calendar index date
6. And does not have original vaccine formulation within 2 months before calendar index date.

By Disease Status, Bivalent

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Has medical and pharmacy enrollment in HealthVerity as of 31 August 2022
2. And is age >=6 months
3. And has continuous medical and pharmacy enrollment for 6 months before the calendar index date
4. And has evidence of 1) moderate/severe immunocompromising condition or separately 2) COVID high-risk condition in a period before the calendar index period (lookback times are dependent on the disease and are provided in variable table below)
5. And has evidence of ≥3 doses of COVID-19 original vaccine formulation before the calendar index date.

For Pregnant Women, Bivalent

Patients must meet all of the following inclusion criteria to be eligible for inclusion in the study:

1. Has at least 6 months of medical and pharmacy enrollment in HealthVerity as of 31 August 2022
2. And is female sex
3. Aged 12-49
4. And has estimated date of pregnancy start date within 9 months before or any point after the calendar entry date (determined using gestational age algorithm)
5. And has evidence of ≥2 doses of COVID-19 original vaccine formulation before the pregnancy start date or 31 August 2022, whichever is latest.
6. And did not receive the bivalent dose prior to pregnancy, if estimated pregnancy start date is after 31 August 2022

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients will be sourced from HealthVerity and include patients who are enrolled in the claims database as well as recorded in contributing states' deidentified vaccine registries. Patients who will be followed for the PCC endpoint must be eligible to receive the licensed/authorized vaccine during the study period.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-09-09 (Actual); Study Completion 2025-09-09 (Actual)

PRIMARY OUTCOMES:
Aim 1: Any PCC-related diagnosis not present before the COVID-19 diagnosis | 30-180 days after COVID-19 diagnosis
  The primary endpoint is any PCC-related diagnosis as defined by Xie et al. (2024, NEJM) that occurs between 30 and 180 days following a COVID-19 diagnosis and was not present before the COVID-19 diagnosis. The primary endpoint will also be stratified by specific organ system / disease domains (cardiovascular; coagulation and hematologic; fatigue; gastrointestinal; kidney; mental health; metabolic; musculoskeletal; neurologic; and, pulmonary). All patients are required to have a diagnosis of COVID-19 (ICD-10-CM code = U07.1) as a predicating event for the subsequent evaluation of a PCC episode. The first 30 days after the diagnosis of COVID-19 will be excluded from the evaluation of a PCC episode as the acute infection period. The evaluation of the PCC episode will begin on Day 30 after the date of acute COVID-19 diagnosis through day 180.
Aim 2: Number of patients with a COVID-19 vaccination | Date of vaccine authorization through the end of the corresponding respiratory season
  Any record of COVID-19 vaccination as recorded in the state immunization registry.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4591059